CLINICAL TRIAL: NCT06355427
Title: The Effect of [18F] F-FAPI PET-CT on Management in Patients With Potentially Resectable Biliary Tract Cancers: Prospective Multicenter Study and Cost-effectivity Analysis
Brief Title: The Effect of [18F] F-FAPI PET-CT on Management in Patients With Proximal Cholangiocarcinoma
Acronym: FAPIChol
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mara Veenstra, MD (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); UMC Utrecht (Other)
Responsible Party: Sponsor-Investigator, Mara Veenstra, MD, Coordinating Investigator, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-507938-24-00
Record Dates: First submitted 2024-03-15; First posted 2024-04-09 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Cholangiocarcinoma
Keywords: FAPI; Cholangiocarcinoma; FAPI PET/CT; Fibroblast Activation Protein Inhibitor; Proximal cholangiocarcinoma; FAPIChol; PET/CT; 18F-FAPI-74
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FAPI PET-CT (Experimental): Participants will undergo additional FAPI PET-CT prior to scheduled surgery.
  Interventions: Drug: [18F]F-FAPI PET-CT

INTERVENTIONS:
Drug: [18F]F-FAPI PET-CT — [18F]F-FAPI PET-CT in addition to regular CT and MRI, prior to participants undergoing surgery

SUMMARY:
Background

Bile duct cancer (cholangiocarcinoma) represents the second most common type of hepatobiliary cancer worldwide with an incidence of 0.35 to 2 per 100.000 annually. Currently, surgical resection is the only curative option. However, patients are not eligible for surgery if the tumor cannot be resected or the cancer has spread. For this group of patients, palliative chemotherapy is the most suited treatment option. To find out if a patient is suited for surgery, CT and MRI are performed. These imaging techniques, however, struggle to correctly identify small cancer spreads that are smaller than 1 cm. Therefore, cancer that has already spread can be found during surgery. In these cases, the tumor cannot be removed and the surgery therefore has not been of any benefit for the patient. These surgeries could be avoided by implementing a diagnostic tool with significantly higher accuracy than those currently used. Single center studies have shown that fibroblast activation protein inhibitor (FAPI) PET-CT is a very promising technique for determining metastases in tumors with prominent desmoplastic reactions, like cholangiocarcinoma. The investigators predict that implementation of preoperative FAPI PET-CT could prevent futile surgery for at least half of patients in whom intra-operative metastasized disease is found using the current work-up.

Patient population

Patients ≥18 years with potentially curable proximal cholangiocarcinoma (perihilar, intrahepatic and gall bladder cholangiocarcinoma) who are planned to undergo surgery based on imaging using CT thorax/abdomen and MRI of the upper abdomen. Exclusion criteria are previous abdominal surgery or chemotherapy, known pregnancy or lactation and indication for FDG PET-CT.

Participation in this study

Participation would mean to undergo FAPI PET-CT prior to the scheduled surgery. This will take up about half a day of the participant's time. Afterwards, participants receive questionnaires about quality of life and use of healthcare services over a period of six months in order for the researchers to be able to calculate the cost-effectiveness of additional FAPI PET-CT.

Risks and benefits of participation

Patients may benefit directly from [18F]F-FAPI PET-CT by allowing for more targeted treatment, possibly avoiding futile surgery and receiving chemotherapy or best clinical support instead, minimizing treatment delay. Avoiding futile surgery will also prevent patients from being exposed to the risks and discomfort associated with surgery: hospital stay, possibility of intraoperative or postoperative complications, postoperative pain and recovery, and mortality.

Potential risks and burdens associated with this study are an extra hospital visit and a time burden of approximately half a day. Risks associated with administering FAPI are (re)bleed and infection. Both risks have a minimal probability of onset and can usually easily be treated. As [18F]F-FAPI is a sub-pharmacologically micro-dosed diagnostic tracer, the risk of allergic reactions is expected to be minimal and no tissue damage is expected. The burden associated with undergoing a PET-CT may be laying still for a certain time, and possible experience of claustrophobia. Possible metastases of the cancer will have to be confirmed when suspicious findings are seen on FAPI PET-CT. This could mean that participants will have to undergo additional testing such as imaging (CT or MRI) or biopsy. Undergoing FAPI PET-CT prior to surgery will result in a surgical delay when compared with the current clinical practice. The investigators do not expect this delay to influence the patient's prognosis. Follow-up will result in a time burden for patients to answer questionnaires on a two-weekly or monthly basis.

DETAILED DESCRIPTION:
Rationale

Bile duct cancer (cholangiocarcinoma) represents the second most common type of hepatobiliary cancer worldwide with an incidence of 0.35 to 2 per 100.000 annually. Currently, surgical resection is the only curative option. However, patients are not eligible for surgery if vascular invasion, distant tumor positive lymph nodes, peritoneal metastases or organ metastases are found on preoperative imaging. For this group of patients, palliative chemotherapy is the most suited treatment option. The preoperative imaging currently includes CT, MRI and FDG PET-CT. In around 29 % of potentially resectable tumors (based on preoperative imaging) metastases are found during subsequent surgery. These explorations could be avoided by implementing a diagnostic tool with significantly higher accuracy than those currently used. Single center studies have shown that fibroblast activation protein inhibitor (FAPI) PET-CT is a very promising technique for determining metastases in tumors with prominent desmoplastic reactions, like cholangiocarcinoma. Our systematic review has shown it is superior to the commonly used FDG PET-CT for this indication. The investigators predict that implementation of preoperative FAPI PET-CT could alter treatment course for at least half (13%) of patients in whom intra-operative metastasized disease is found using the current work-up.

Objective

The primary aim of this study is to assess whether preoperative [18F]F-FAPI PET-CT in addition to standard preoperative imaging can successfully identify metastasized disease and change treatment plan in patients with potentially resectable proximal bile duct cancer (intrahepatic, perihilar and gall bladder cholangiocarcinoma). This study also aims to evaluate if adding [18F]F-FAPI PET-CT to preoperative imaging is cost-effective.

Main trial endpoints

The main endpoint is the diagnostic accuracy (sensitivity, specificity, positive predictive value, negative predictive value) of [18F]F-FAPI PET-CT.

Secondary trial endpoints

* Diagnostic accuracy of [18F]F-FAPI PET-CT per abdominal region and per lesion
* The number of additional significant findings on [18F]F-FAPI PET-CT
* Change of treatment: true change and virtual change
* The number of times readers' conclusions differed and why
* Cost-effectiveness analysis, budget impact analysis (BIA), sector costs, societal costs, health-related quality of life (HRQoL)
* The number of additional significant findings on [18F]F-FAPI PET-CT
* Number of days between date of first imaging (CT/MRI) and starting date of chemotherapy, palliative therapy or surgical resection
* The incidence and severity of AEs and SAEs according to CTCAEv5
* VOI, TTP, K1 and k2, SUV and TBR (in a subgroup of patients)

Trial design

Prospective multicenter observational cohort study, expected total duration 4 years. Participants will be participating for at least six months.

Trial population

Patients ≥18 years with potentially curable proximal cholangiocarcinoma (perihilar, intrahepatic and gall bladder cholangiocarcinoma) who are planned to undergo surgery based on imaging using CT thorax/abdomen and MRI of the upper abdomen. Exclusion criteria are previous abdominal surgery or chemotherapy, known pregnancy or lactation and indication for FDG PET-CT.

Interventions

If patients are deemed eligible for surgery (laparoscopy or laparotomy) by the weekly organ-specific multidisciplinary team (MDT) including an abdominal nuclear medicine specialist, radiologist, surgeon, gastroenterologist/hepatologist, oncologist and, optionally, pathologist, patients will be asked to participate in the study. After inclusion, patients will receive additional [18F]F-FAPI PET-CT. Patients who underwent [18F]F-FAPI PET-CT will undergo follow-up for at least six months, if clinically advisable. Follow-up includes information regarding additional imaging, surgery or complications. To determine cost-effectiveness, patients' medical consumption will be elicited using two questionnaires. Patients will be asked to fill out the 'institute for Medical Technology Assessment (iMTA) Medical Consumption Questionnaire (iMCQ)' at three and six months after their initial CT/MRI imaging (before [18F]F-FAPI PET-CT or surgery). Patients will also be asked to fill out the European Organisation for Research and Treatment of Cancer (EORTC) group's QLQ-C30 and QLQ-BIL21 questionnaires and the EuroQol (EQ) Group's EQ-5D-5L questionnaire once every two weeks during the first two months after [18F]F-FAPI PET-CT and then once every four weeks until six months follow-up.

Risks and benefits

Patients may benefit directly from [18F]F-FAPI PET-CT by allowing for more targeted treatment, possibly avoiding futile surgery and receiving chemotherapy or best clinical support instead, minimizing treatment delay. Avoiding futile surgery will also prevent patients from being exposed to the risks and discomfort associated with surgery: hospital stay, possibility of intraoperative or postoperative complications, postoperative pain and recovery, and mortality.

Potential risks and burdens associated with this study are an extra site visit and a time burden of approximately half a day. Risks associated with vena puncture are (re)bleed and infection. Both risks have a minimal probability of onset, and when anticipated upon, are not expected to have significant clinical consequences. Risks associated with the administration of the study agent are allergic reactions and radiation burden. [18F]F-FAPI is a sub-pharmacologically micro-dosed diagnostic tracer, which is why the risk of allergic reactions is expected to be minimal and no tissue damage is expected. The burden associated with undergoing a PET-CT may be laying still for a certain time, and possible experience of claustrophobia. Metastases will have to be confirmed when suspicious findings are seen on [18F]F-FAPI PET-CT. This could mean subjects will have to undergo additional testing such as imaging (CT or MRI) or biopsy. If these additional tests are negative for metastases, the subject's exploratory surgery will have been needlessly delayed. Having to undergo [18F]F-FAPI PET-CT prior to surgery will also result in a surgical delay when compared with the current clinical practice. The investigators do not expect this delay to influence the subject's prognosis. Follow-up will result in a time burden for patients to answer questionnaires on a two-weekly or monthly basis.

ELIGIBILITY:
Inclusion Criteria:

* Patient is scheduled for explorative laparoscopy or laparotomy for suspicion of proximal cholangiocarcinoma (perihilar, intrahepatic and gall bladder cholangiocarcinoma)
* Tumor is regarded as resectable based on preoperative CT and MRI
* Patient is 18 years or older and is able to give informed consent

Exclusion Criteria:

* Previous abdominal surgery or chemotherapy
* Patient had FDG PET-CT in addition to preoperative CT and MRI
* Contra-indication for performing PET-CT
* Indication for FDG PET-CT
* Pregnancy or lactation, for the latter, temporary discontinuation may be considered.
* Known allergic reaction to therapeutic radiopharmaceuticals
* Inability to lie still on the back for the duration of PET-CT
* Impaired renal function, defined as eGFR (MDRD) <25 ml/min/1,73 m2. An exception can be made in consultation with the treating physician.
* Any (other) condition, disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that may affect the interpretation of the results, or which might contribute substantially to the patient's experience of study burden (such as non-suppressible claustrophobia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of [18F]F-FAPI PET-CT | Six months following PET-CT
  Diagnostic accuracy will be expressed using sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV)

SECONDARY OUTCOMES:
Change of treatment | Within one month following PET-CT
  Change of treatment is based on a combination of true change during work-up and virtual change based on [18F]F-FAPI PET-CT findings, with proof during further exploration (laparoscopy or laparotomy), resection or follow-up. True change is defined as a positive finding that changes the intent of treatment, i.e. no explorative laparoscopy/laparotomy and no resection. Virtual change of therapy is defined as a positive finding with FAPI PET-CT, which should preclude explorative laparoscopy and resection but where the latter is still performed.
Cost-effectiveness | Six months following PET-CT
  Determining the value of introducing [18F]F-FAPI PET-CT in terms of quality-adjusted life years (QALY) and costs compared to the current standard of care (SoC).
Number of additional significant findings using [18F]F-FAPI PET-CT | Within one week after PET-CT
  Additional significant findings include other primary tumors (albeit benign or malignant) and other relevant findings such as infectious and inflammatory processes.
Number of times nuclear medicine specialists' [18F]F-FAPI PET-CT conclusions differed from one another | Within one week after PET-CT
  To assess the inter-reader variability between nuclear medicine specialists. Consensus regarding the presence of metastases, lymph node involvement, and the location of possible metastases and/or suspicious lymph nodes will be assessed.
Number of lesions found on [18F]F-FAPI PET-CT | Within one week after PET-CT
  The amount of suspicious findings on [18F]F-FAPI PET-CT
Number of days between [18F]F-FAPI PET-CT and exploratory surgery | Six months following PET-CT
  Differences in treatment delay between patients with and without significant findings on [18F]F-FAPI PET-CT will be assessed. Treatment delay is defined as the time in days from the first multidisciplinary team meeting to exploratory surgery.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Six months following PET-CT
  Measured by the incidence and severity of AEs and SAEs according to CTCAE v5.0
Number of participants in which dynamic [18F]F-FAPI PET-CT followed by conventional [18F]F-FAPI PET-CT was able to distinguish benign lesions from malignant lesions | Six months following PET-CT
  Subgroup analysis. As part of the subgroup analysis participants undergo dynamic [18F]F-FAPI PET-CT followed by conventional PET-CT at one hour post-injection.
Change in volume of interest (cm3) using dynamic [18F]F-FAPI PET-CT | Within one week after PET-CT
  Subgroup analysis. As part of the subgroup analysis participants undergo dynamic [18F]F-FAPI PET-CT followed by conventional PET-CT at one hour post-injection.
Difference in SUVmax between dynamic and conventional [18F]F-FAPI PET-CT | Within one week after PET-CT
  Subgroup analysis. As part of the subgroup analysis participants undergo dynamic [18F]F-FAPI PET-CT followed by conventional PET-CT at one hour post-injection.
Difference in SUVmean between dynamic and conventional [18F]F-FAPI PET-CT | Within one week after PET-CT
  Subgroup analysis. As part of the subgroup analysis participants undergo dynamic [18F]F-FAPI PET-CT followed by conventional PET-CT at one hour post-injection.
Difference in transport rate (k1 to k2) on dynamic [18F]F-FAPI PET-CT between participants with malignant lesions and particpants with benign lesions | Six months following PET-CT
  Subgroup analysis. As part of the subgroup analysis participants undergo dynamic [18F]F-FAPI PET-CT followed by conventional PET-CT at one hour post-injection.

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Amsterdam UMC, Amsterdam
  - Erasmus MC, Rotterdam
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided